CLINICAL TRIAL: NCT06823141
Title: Effect of Virtual Reality Immersion on Patient's Anxiety During Pre-oxygenation Before General Anaesthesia: a Pilot Study
Brief Title: Effect of Virtual Reality Immersion on Patient's Anxiety During Pre-oxygenation Before General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Schlotterbeck Hervé, Medical Doctor, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID 2024-02157
Record Dates: First submitted 2025-01-23; First posted 2025-02-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Pre-oxygenation; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality arm (Experimental)
  Interventions: Device: Virtual reality immersion

INTERVENTIONS:
Device: Virtual reality immersion — The study intervention, defined by the use of a virtual reality, exclusively takes place during the pre-oxygenation period where the patient is exposed to a virtual reality immersion scenario.

SUMMARY:
The goal of this clinical trial is to learn if the use of virtual reality immersion during pre-oxygenation before general anesthesia could be feasible and beneficial for the patient. The main questions it aims to answer are:

Does virtual reality immersion during pre-oxygenation reduce patient's anxiety? Does it impact patient's and anaesthetist's comfort? Is this technique easy to implement?

ELIGIBILITY:
Inclusion Criteria:

* All non-ambulatory patients undergoing elective surgery or procedure under general anaesthesia with intravenous induction
* Minimal age of 18 year old
* Able to give informed consent for the study as documented by signature

Exclusion Criteria:

* Lacking capacity or ability to complete the consent form and/or questionnaire and interview method and/or incapacity to respond to the required obligations linked to the study protocol (assessed by the operator)
* Known cognitive dysfunction, previous history of neurological/psychiatric disease like epilepsy
* Depression or anxiety under treatment
* Non-Italian speaking patients
* Anticipated difficult airway management
* Injuries to the head/face that would prohibit wearing headsets
* Active nasal bleeding or occlusion, nasal abnormality or recent nasal trauma, recent nasal surgery, significant raised intracranial pressure and base of skull fractures
* Any pre-operative premedication, including pharmacological premedication
* Rapid sequence induction
* Haemodynamic instability
* Infectious skin conditions on the head/face
* Undrained pneumothorax
* Contact isolation due to bacteria and viruses
* Symptoms of vertigo or motion sickness
* Reduced visual or auditory acuity
* BMI > 35 kg/m2
* Pregnancy
* Claustrophobia
* Pre-existing hypoxemia (baseline oxygen saturation < 92% when breathing room air)
* Need for an arterial line before general anaesthesia induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Patient's Anxiety during pre-oxygenation | 4 min after the beginning of pre-oxygenation.
  Anxiety will be assessed with the Visual Analogue Scale for Anxiety (VASA) scale ranging from 0 to 10 (0 corresponds to the lowest level of anxiety and 10 to maximal level of anxiety).

SECONDARY OUTCOMES:
Change in patient's anxiety over time | The four time points are: in the ward on the day of surgery, in the theater once the patient is monitored and before pre-oxygenation, 4 min after the beginning of pre-oxygenation, in the ward at least two hours after the end of surgery.
  Change in Visual Analogue Scale for anxiety (VASA) between 4 time points. VASA scale ranges from 0 to 10 with 10 corresponding to the highest level of anxiety.
Success rate in recruiting patients to participate to the study | During study recruitment.
  Rate of patients accepting to participate to the study. The number of patients accepting to participate will be descrided in percent (%) with the denominator beeing the sum of patients who accepted and refused to participate to the study.
Completed pre-oxygenation with virtual reality headset | From the beginning to the end of the pre-oxygenation period.
  Rate of patient who completed pre-oxygenation with the virtual reality headset. The rate of patient who completed the pre-oxygenation with the virtual reality headset will be measured in percent (%).
Anxiety evaluation with the Amsterdam Preoperative Anxiety and Information scale (APAIS) score | At two times: on the day of surgery while the patient is still in the ward and after entry in the OR up to the beginning of pre-oxygenation.
  The APAIS score is a validated score to evaluate anxiety in the preoperative context. It ranges from 6 to 30 with the highest score corresponding to a high level of anxiety.
Change in blood pressure over time | The four time points are: in the ward on the day of surgery, the first blood pressure measured in theater, at the beginning of the pre-oxygenation and at the end of the pre-oxygenation (just before the beginning of the general anaesthesia induction)
  Variation of blood pressure (systolic arterial pressure, diastolic arterial pressure, mean arterial pressure) between four time points.
Change in oxygen saturation over time | The four time points are: in the ward on the day of surgery, the first oxygen saturation measured in theater, at the beginning of the pre-oxygenation and at the end of the pre-oxygenation (just before the beginning of the general anaesthesia induction)
  Variation of oxygen saturation measured with finger pulsoxymeter between four time points.
Change in heart rate over time | The four time points are: in the ward on the day of surgery, the first heart rate measured in theater, at the beginning of the pre-oxygenation and at the end of the pre-oxygenation (just before the beginning of the general anaesthesia induction)
  Variation of heart rate measured between four time points.
Patient's comfort during pre-oxygenation | During pre-oxygenation (at 2 minutes after pre-oxygenation initiation).
  Patient will be asked it's level of comfort during pre-oxygenation with a Likert scale ranging from 0 to 10 (with 0 corresponding to the maximum comfort and 10 to the minimal comfort).
Incidence of cybersickness | From the beginning to the end of the pre-oxygenation period.
  Incidence of cybersickness during the pre-oxygenation period in percent (%).
Comfort of the anesthetic team during pre-oxygenation | From the beginning to the end of the pre-oxygenation period.
  Evaluation of the involved anesthetic team comfort regarding the pre-oxygenation technique with a Likert scale ranging from 1 to 5 (1 corresponding to the lowest level of comfort and 5 to the highest level of comfort).
Perceived comfort of the patient during pre-oxygenation | From the beginning to the end of the pre-oxygenation period.
  Perceived comfort of the patient during pre-oxygenation by the involved anesthetist team with a Likert scale ranging from 1 to 5 (1 beeing the lowest level of comfort and 5 beeing the highest level of comfort).
Wake up quality test | From the beginning of the awakening after general anesthesia to the removal of the airway device.
  Wake up quality test with a 3-point scale (good, satisfactory, poor).
Patient's satisfaction regarding the pre-oxygenation period | From 2 hours after the end of anesthesia to the first day after surgery.
  Evaluation of patient's satisfaction regarding the pre-oxygenation technique with a 5-point Likert scale (1 beeing the lowest level of satisfaction and 5 the highest level of satisfaction)
Qualitative post-operative survey regarding patient's experience during pre-oxygenation | From 2 hours after the end of anesthesia to the first day after surgery.
  Qualitative post-operative survey with questions about patient's experience during pre-oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Cardiocentro, Lugano, Canton Ticino, Switzerland